CLINICAL TRIAL: NCT01382394
Title: Impact of Clinical, Demographic and Laboratory Variables on Brain Natriuretic Peptide Levels
Status: Withdrawn | Type: Observational
Why Stopped: No Patients were recruited during the study period
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Rambam Medical Center, Zaher S. Azzam M.D.
Other Study IDs: 0459-09-RMB
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Sepsis; Heart Failure
Keywords: Sepsis; heart failure; BNP; IL-6; Procalcitonin; Prognosis
MeSH Terms: conditions — Sepsis; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sepsis Group, Heart failure group: The first group will include 60 patients with the diagnosis of acute decompensated heart failure.
  The second group will include 60 patients with the diagnosis of sepsis.

SUMMARY:
Brain natriuretic peptide (BNP) is involved in the regulation of blood pressure and fluid volume. It is used for the early diagnosis of heart failure (HF) in patients presenting to the emergency room with dyspnea. Interleukin-6 (IL-6) is a cytokine marker of inflammation that exhibits significant prognostic value in predicting severity and outcome of sepsis. Recently, it was suggested that inflammatory cytokines play an important role in the development of heart failure. Procalcitonin (PCT) is a propeptide of calcitonin which is normally produced in the C-cells of the thyroid glands. Although physiologic levels of PCT remain very low, a dramatic increase in serum PCT levels is observed during severe systemic infections. These properties make procalcitonin less useful for the diagnosis of simple infections but a very promising marker of severe infections especially in the critical care setting.

To investigate the co-relation between BNP, IL-6 and procalcitonin in two groups of patients; those presenting with the diagnosis of decompensated heart failure and in patients presenting with the diagnosis of sepsis without cardiovascular or hemodynamic dysfunction.

DETAILED DESCRIPTION:
Brain natriuretic peptide (BNP), forms together with atrial natriuretic peptide (ANP) a peptide family involved in the regulation of blood pressure and fluid volume. It is used for the early diagnosis of heart failure (HF) in patients presenting to the emergency room with dyspnea. Additionally, in patients with chronic HF and acute and chronic coronary syndrome, BNP is a marker of unfavorable prognosis, being associated with increased mortality.

Recently, elevated BNP levels have been measured in patients with septic shock and have been attributed to myocardial dysfunction due to sepsis. Because BNP synthesis is also induced by endotoxin and inflammatory mediators, the mechanisms leading to elevated BNP levels in patients with sepsis remain unclear.

Interleukin-6 (IL-6) is a cytokine marker of inflammation that exhibits significant prognostic value in predicting severity and outcome of sepsis, since it is considered to play a key role in the pathogenesis of sepsis. Accumulating evidence suggests that inflammatory cytokines play an important role in the development of heart failure. In particular, studies using genetically engineered animal models have demonstrated the critical role of the gp130-dependent cardiomyocyte survival pathway in the transition to heart failure. However, the significance of gp130 for patients with CHF has not been fully assessed. Previous clinical studies showed that the plasma level of IL-6 is elevated in patients with advanced CHF and that such high levels are associated with a poor prognosis for CHF patients.

Procalcitonin (PCT) is a propeptide of calcitonin which is normally produced in the C-cells of the thyroid glands. Although physiologic levels of PCT remain very low, a dramatic increase in serum PCT levels is observed during severe systemic infections. It is not infection per se but infection accompanied by severe systemic reactions or poor organ perfusion that increases procalcitonin levels. These properties make procalcitonin less useful for the diagnosis of simple infections but a very promising marker of severe infections especially in the critical care setting.

Few studies have investigated the role of procalcitonin in patients with acute heart failure, although there was a slightly increased level of procalcitonin in patients with severe acute heart failure, the results were not conclusive. These results support the hypothesis that inflammatory process has a role in heart failure.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with decompensated heart failure (N-60).
* 2) Patients with sepsis (N-60).

Exclusion Criteria:

* 1) Patients who are under the age of 18 years
* 2) pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed at Rambam Medical Center, Israel. Patients admitted to the department of internal medicine will be divided to two groups
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaher S Azzam, MD, Study Chair — Head Of Internal Medicine "B"
Locations (1):
- Internal Medicine "B", Rambam Medical center, Haifa, Israel